CLINICAL TRIAL: NCT06201208
Title: The Effect on Well-Being, Self-Transcendence, Self-Reflection and Insight of the Self-Transcendence Facilitation Psychoeducational Program Applied to Mothers of Children With Special Needs
Brief Title: Self-Transcendence Facilitation Psychoeducational Program Applied to Mothers of Children With Special Needs
Acronym: STFacilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, YELDA KUBLAY, Lecturer, Akdeniz University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 70904504/516
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Mothers; Special Needs Children; Psychoeducation; Well-being
Keywords: well being; self-reflection; insight; mother; special needs children; self-transdence theory; psychoeducation program; psychiatric nursing

STUDY DESIGN:
Intervention Model Description: This study is a non-randomized experimental study with pre-test, post-test, follow-up and control groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ST-Facilitation Psychoeducation Program Group (Experimental): The ST-Facilitation Psychoeducation Program is planned for mothers in the intervention group as an 80-minute session (40-minute session + 20-minute break + 40-minute session) once a week for six weeks, in groups of two to four participants.
  Interventions: Behavioral: The ST-Facilitation Psychoeducation Program
- Control Group (No Intervention): No action will be taken by the researcher during the research. Only data collection will be carried out. At the end of the research, ST-Facilitation Psychoeducation Program will be applied ethically.

INTERVENTIONS:
Behavioral: The ST-Facilitation Psychoeducation Program — One of the important roles of the psychiatric nurse, who helps healthy/sick individuals and their families to improve their mental health, prevent and cope with diseases, is their educational role. The psychiatric nurse determines the psychosocial care needs of the patient and his family and plans, implements and evaluates psychoeducational interventions, which are an evidence-based practice, to meet these needs.
  Psychiatric nurses can benefit from existing programs when developing a psychoeducation program, or they can be advised to create programs that include educational and psychosocial goals based on theory specific to the problems of the relevant population. The theoretical basis is of great importance when planning a psychoeducation program. In this study, the psychoeducation program was based on the Self-Transcendence Theory of Pamela G. Reed, a psychiatric nurse.
  Arms: The ST-Facilitation Psychoeducation Program Group

SUMMARY:
This study aimed to determine the effect of the Facilitating Self-Transcendence Psychoeducation Program, which will be applied to mothers of children with special needs, on well-being, self-transcendence, self-reflection, and insight.

DETAILED DESCRIPTION:
This study aimed to determine the effect of the Facilitating Self-Transcendence Psychoeducation Program, which will be applied to mothers of children with special needs, on well-being, self-transcendence, self-reflection and insight.

This study is a non-randomized experimental study with pre-test, post-test, follow-up and control groups. A 2x3 split-plot factorial design will be used as the research design. In this design, the first factor shows independent interventional procedure groups, and the second factor shows repeated measurements of the dependent variable (pre-test, post-test and follow-up). Considering the theoretical basis of psychoeducational programs, the follow-up period in this study was planned to be eight weeks after the last session.

The study will be carried out between February 2024 and July 2024. The sample of the study will consist of mothers of children with special needs between the ages of 0-11 who are registered in a special education and rehabilitation center in Kumluca. 30 mothers will be included in the intervention group and 30 mothers in the control group. The ST-Facilitation psychoeducation program is planned for mothers in the intervention group as an 80-minute session (40-minute session + 20-minute break + 40-minute session) once a week for six weeks, in groups of two to four people. Data will be collected using the Personal Information Form, Self-Transcendence Scale, Warwick-Edinburgh Mental Well-Being Scale and Self-reflection and Insight Scale.

ELIGIBILITY:
Inclusion Criteria:

Volunteering to participate in research No cognitive disabilities such as reading, writing, communication and understanding No possibility of leaving the region during the research. Being a mother of a child with special needs between the ages of 0-11

Exclusion Criteria:

Continuing psychiatric treatment during the period when the study was conducted Involvement in another psychosocial intervention that is likely to influence the research outcome.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Well-Being Scale | 6 months
  Warwick-Edinburgh Mental Well-Being Scale consists of 14 items and a single dimension. The scale is five-point Likert type. Scoring of the scale is as follows: 1 = strongly disagree, 2 = disagree, 3 = somewhat agree, 4 = agree, 5 = completely agree. All items of the scale are positive and there is no cut-off score. The minimum score from the scale is 14 and the maximum score is 70. High scores from the scale indicate high mental well-being.
Self-Transcendence Scale | 6 months
  Self-Transcendence Scale is a unidimensional scale consisting of 15 items. The scale is a four-point Likert type. Scoring of the scale is as follows: 1 = not at all, 2 = very little, 3 = quite a bit, 4 = very much. All items of the scale are positive and there is no cut-off score. A minimum of 15 and a maximum of 60 points are obtained from the scale. Increasing scores from the scale are evaluated as increasing self-transcendence.
Self-reflection and Insight Scale | 6 months
  The scale consists of 20 items and two factors. These factors are "self-reflection" and "insight"; The "self-reflection" factor has two sub-dimensions: being dependent on self-reflection and needing self-reflection. There are 8 items in the "insight" factor of the scale and 12 items in the "self-reflection" factor. The scale is a six-point Likert type. Scoring of the scale is 1 = strongly disagree, 2 = disagree, 3 = partially disagree, 4 = partially agree, 5 = agree, 6 = strongly agree. Items that require reverse scoring are items 1, 2, 4, 8, 9, 11, 13, 14 and 17. In reverse scoring, a score of "1" becomes "6"; "2" becomes "5"; "3" becomes "4" and vice versa. No scaling or scale conversion is required other than basic reverse scoring. A minimum of 20 and a maximum of 120 points are obtained from the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Kumluca, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to preserve the originality of the research, it is not intended to be shared until the research is completed and reaches the publication stage.